CLINICAL TRIAL: NCT03508492
Title: Comparative Study to Asses the Satisfaction With Tinted Chlorhexidine Applicators (Chloraprep® and Nex Clorex 2%)
Brief Title: Surgeons' Satisfaction With Two Types of Tinted Chlorhexidine Applicators (Chloraprep® and Nex Clorex 2%)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cristina Fernandez Perez (Other)
Responsible Party: Sponsor-Investigator, Cristina Fernandez Perez, Head of Preventive and Public Health Department, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CA-IQZ
Record Dates: First submitted 2018-04-05; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Satisfaction; Product Quality
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Knee surgeons (Active Comparator): Four knee surgeons
  Interventions: Other: Surgical tinted Chloraprep® applicators; Other: Surgical tinted Nex Clorex 2% applicators
- Hip surgeons (Active Comparator): Six hip surgeons
  Interventions: Other: Surgical tinted Chloraprep® applicators; Other: Surgical tinted Nex Clorex 2% applicators
- Cardiac surgeons (Active Comparator): 6 cardiac surgeons
  Interventions: Other: Surgical tinted Chloraprep® applicators; Other: Surgical tinted Nex Clorex 2% applicators
- Colon surgeons (Active Comparator): 6 colon surgeons
  Interventions: Other: Surgical tinted Chloraprep® applicators; Other: Surgical tinted Nex Clorex 2% applicators

INTERVENTIONS:
Other: Surgical tinted Chloraprep® applicators — We randomized knee, hip, cardiac and colon surgeons making them using two applicators of each brand in four of theirs surgeries. Randomization will be carried out in blocks of four for each surgeon.
Other: Surgical tinted Nex Clorex 2% applicators — We randomized knee, hip, cardiac and colon surgeons making them using two applicators of each brand in four of theirs surgeries. Randomization will be carried out in blocks of four for each surgeon.

SUMMARY:
The development of surgical site infections (SSI) in clean-contaminated surgery is regarded as being preventable. Known to be effective in the prevention of surgical site infection are the adequate sterilization of the surgical instruments, asepsis during operation, antibiotic prophylaxis where indicated, and certainly the preparation of the skin at the incision site. During the last decades the use of alcoholic chlorhexidine has replaced povidone iodine for preoperative skin preparation. In order to improve the way alcoholic chlorhexidine is applied, pharmaceutical industry has developed new applicators.

This randomized study was conducted to know the surgeons' satisfaction within the use of two tinted applicators: Chloraprep® and Nex Clorex 2%

ELIGIBILITY:
Inclusion Criteria:

* Volunteer surgeons from colon, cardiac, knee and hip surgical departments. Once surgeon has enrolled the study, patients will be selected if they have hospital admission with scheduled surgery and have signed informed consent

Exclusion Criteria:

* Urgent surgeries
* Outpatient surgery
* Surgical complex cures
* Mixed interventions: exploratory or sequential
* Unscheduled surgeries
* Rejection of participation
* Chlorhexidine or isopropyl alcohol hypersensibility patients
* If any patients changed its mind after signing the informed consent will be removed from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Surgeon's global satisfaction with the applicators. | Intraoperative
  Using an analog visual scale we will record the total score, over a maximum of 80 points, that assess the following quality aspects of the applicators:
  * Satisfaction with the presentation of the product
  * Satisfaction with the simplicity of activation
  * Satisfaction with the mix of the different components of the product
  * Satisfaction with the comfort of product use
  * Satisfaction with the surface covered by an applicator
  * Satisfaction with the shape of the applicator for painting areas of difficult access
  * Satisfaction with the drying time of the product
  * Satisfaction with the area delimited with the use of the product
Qualities of each applicators | Intraoperative
  Using an analog visual scale, were one end represents "totally disagree" and the other "totally agree" (0-10 points), we will record the score of each of the following quality aspects of the applicators:
  * Satisfaction with the presentation of the product
  * Satisfaction with the simplicity of activation
  * Satisfaction with the mix of the different components of the product
  * Satisfaction with the comfort of product use
  * Satisfaction with the surface covered by an applicator
  * Satisfaction with the shape of the applicator for painting areas of difficult access
  * Satisfaction with the drying time of the product
  * Satisfaction with the area delimited with the use of the product

SECONDARY OUTCOMES:
Costs of using the applicators | Through study completion, an average of 3 months
Adhesion to preoperative measures to avoid surgical site infections (SSI) | Through study completion, an average of 3 months
  Analyze the verification check list for surgical site infection preoperative prevention. This check list has been provided by the Preventive Medicine, Public Health and Hygiene Spanish Society as part of the Zero Surgical Site Infection Protocol.
  This verification check list includes indicators of:
  * Antibiotic prophylaxis
  * Intraoperative Alcoholic Chlorhexidine application
  * Hair removal from the surgical site
  * Normotherapy
  * Glycemic control
Surgical site infection incidence | During the first 30 to 90 days after surgery, according to the SSI prevention protocol